CLINICAL TRIAL: NCT04632199
Title: A Phase I, Open Label, Study to Assess Safety, Tolerability, Biodistribution, Radiation Dosimetry and SPECT/CT Imaging Characteristics of Intravenous 111In-IPN01087 in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma or Colorectal Cancer.
Brief Title: Study to Assess the Safety and Efficacy of Intravenous Injection of the Imaging Agent 111In-IPN01087 in Patients With Locally Advanced or Metastatic Pancreatic or Colorectal Cancer.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision not related to any safety or tolerability concern
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D-FR-01087-002; 2019-002882-37 (EudraCT Number)
Record Dates: First submitted 2020-10-23; First posted 2020-11-17 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 111In-IPN01087 Low dose (Experimental): Single intravenous injection of 220 MBq 111In-IPN01087 with a low mass dose of IPN01087
  Interventions: Drug: 111In-IPN01087 Low dose
- 111In-IPN01087 High dose (Experimental): Single intravenous injection of 220 MBq 111In-IPN01087 with a high mass dose of IPN01087
  Interventions: Drug: 111In-IPN01087 High dose

INTERVENTIONS:
Drug: 111In-IPN01087 Low dose — Administered once via slow intravenous injection.
  Arms: 111In-IPN01087 Low dose
Drug: 111In-IPN01087 High dose — Administered once via slow intravenous injection.
  Arms: 111In-IPN01087 High dose

SUMMARY:
111Indium-labelled IPN01087 (111In-IPN01087) is developed as a radioactive diagnostic imaging agent in patients with colorectal or pancreatic cancer. It is used with single-photon emission computed tomography (SPECT) for the identification of tumours that overexpress the neurotensin receptor-1 (NTSR1). The purpose of this study is to assess how well 111In-IPN01087 is tolerated and what the most suitable amount to be injected is to obtain good quality images. The study will also look at how 111In-IPN01087 is distributed throughout the body and what the optimal time for doing the scans will be after it has been given as a single intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form prior to all study procedures.
* Male or female patients ≥18 years.
* Histologically confirmed locally advanced or metastatic Pancreatic ductal adenocarcinoma (PDAC) or Colorectal cancer (CRC), not amenable to treatment with curative intent.
* At least one lesion identified by CT or MRI as being ≥2 cm in the longest diameter on axial plane, which has not been previously treated with external beam radiation.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2.
* Estimated life expectancy >3 months.
* Clinically acceptable medical history, physical examination and vital signs findings during the screening period
* Adequate organ function as evidence by: Leukocytes ≥2000/μL, Absolute neutrophil count ≥750/μL, Platelets ≥75,000/μL, Haemoglobin ≥10 g/dL, Total serum bilirubin ≤1.5×upper limit of normal range (or in case of hepatic metastases ≤2.5 x upper limit of normal range), Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3×upper limit of normal range (or in case of hepatic metastases ≤5 x upper limit of normal range), Estimated glomerular filtration rate ≥50 mL/min.
* Willing and able to comply with study restrictions, including remaining at the clinic for the required time during the study period, and willing to return to the clinic for the follow-up evaluation, as specified in the protocol.
* For women of childbearing potential (neither surgically sterile nor post-menopausal defined as no menses for 12 months without an alternative medical cause), a negative highly sensitive pregnancy test must be documented at the screening visit (serum test).
* Female patients of childbearing potential (not surgically sterile or post-menopause defined as no menses for 12 months without an alternative medical cause) must use a medically accepted highly effective method of contraception and must agree to use this method for the duration of the study (from screening until 6 months after administration of 111In-IPN01087).
* Male patients must agree to use a condom for the duration of the study and for at least 90 days after administration of 111In-IPN01087.
* Male patients with female partners of childbearing potential must use a medically accepted highly effective method of contraception and must agree to use this method for the duration of the study and for at least 90 days after administration of 111In-IPN01087.

Exclusion Criteria:

* Known allergy to the investigational imaging product (IIP) or its excipients administered in this study.
* Any newly commenced licensed or investigational anti-cancer therapy within 30 days prior to IIP administration. Therapies started more than 30 days prior to IIP administration can be continued, provided patients have adequate organ function as per inclusion criteria.
* Receiving, or scheduled to receive, another IIP from 1 month before screening to 1 week after administration of 111In-IPN01087.
* Administration of any radiopharmaceutical within eight half lives of that radionuclide before IIP administration.
* Any unresolved NCI-CTCAE Grade 2 or higher (except alopecia or where Grade 3 is permissible as per the inclusion criteria)
* Any condition that precludes adequate SPECT and/or CT imaging, e.g. patients unable to lie still for the entire imaging time, or metal prosthetics which interfere with CT (hip and knee prosthetics are acceptable).
* Clinically significant abnormalities on ECG at screening
* Any uncontrolled significant medical, psychiatric or surgical condition or laboratory finding that would pose a risk to patient safety, or interfere with study participation, or interpretation of individual patient results.
* Pregnancy, lactation, or breastfeeding.
* Unable to understand the nature, scope and possible consequences of the study, in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-12 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent adverse events | From baseline until the end of study (12 months)
  Safety and Tolerability

SECONDARY OUTCOMES:
Whole body biodistribution of 111In-IPN01087 using whole body planar imaging | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Maximum uptake by source region and the entire body | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Time-integrated activity coefficients by source region and the entire body | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Absorbed Radiation doses per organ | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Specific absorbed radiation doses per organ | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Organs receiving the highest radiation dose. | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Normalized whole body effective dose | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Total effective dose | Day 1 (30 minutes and 6 hours post-dose), Day 2, Day 3 and Day 4
Optimal imaging time window assessed as maximum tumour contrast on single photon emission computed tomography/computed tomography (SPECT/CT) imaging at all available timepoints post injection | Day 1 (6 hours post-dose), Day 2, Day 3 and Day 4
Time for maximal activity in blood | Day 1 (pre-dose, immediately after the end of the 111In-IPN01087 injection (Time 0), 30 minutes, 2 hours, 4 hours and 6 hours post-dose), Day 2, Day 3 and Day 4
Area under the time-activity curve from time 0 to the time of the last quantifiable concentration | Day 1 (pre-dose, immediately after the end of the 111In-IPN01087 injection (Time 0), 30 minutes, 2 hours, 4 hours and 6 hours post-dose), Day 2, Day 3 and Day 4
Apparent terminal elimination half life | Day 1 (pre-dose, immediately after the end of the 111In-IPN01087 injection (Time 0), 30 minutes, 2 hours, 4 hours and 6 hours post-dose), Day 2, Day 3 and Day 4
Cumulative amount of 111In-IPN01087 excreted in the urine over 48 hours | From the time of the 111In-IPN01087 injection to 6 hours, from 6 hours to 24 hours and from 24 hours to 48 hours
Fraction of the administered 111In-IPN01087 excreted in urine over 48 hours | From the time of the 111In-IPN01087 injection to 6 hours, from 6 hours to 24 hours and from 24 hours to 48 hours
Renal clearance of 111In-IPN01087 | From the time of the 111In-IPN01087 injection to 48 hours
Optimal injected radioactivity range | Day 1 (6 hours post-dose), Day 2, Day 3 and Day 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (5):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- France (3):
  - Centre Léon Bérard, Léon
  - CHRU de Nancy - Hôpital de Brabois, Nancy
  - CHU de Nantes - Hôpital Hôtel Dieu, Nantes

IPD SHARING:
Plan to Share IPD: No